CLINICAL TRIAL: NCT04671316
Title: A Open-Label, Randomized, 6-sequence, 3-period, Fasting Condition, Singledose, Per Oral, Cross-over Study to Evaluate the Bioequivalence Between "DA-5209 60mg Tab" and "Lixiana 60mg Tab" in Healthy Volunteers
Brief Title: Bioequivalence Study Between "DA-5209 Tab" and "Lixiana Tab"
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DDS20-035BE
Record Dates: First submitted 2020-11-23; First posted 2020-12-17 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Crossover Assignment single-dose, 6-sequence, 3-period Bioequivalence Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- T1T2R (Experimental): Period I: T1, "DA-5209 60mg" without water Period II: T2, "DA-5209 60mg" with 150mL water Period III: R, "Lixiana 60mg" with 150mL water
  Interventions: Drug: DA-5209 60mg Tab; Drug: Lixiana 60mg Tab
- T1RT2 (Experimental): Period I: T1, "DA-5209 60mg" without water Period II: R, "Lixiana 60mg" with 150mL water Period III: T2, "DA-5209 60mg" with 150mL water
  Interventions: Drug: DA-5209 60mg Tab; Drug: Lixiana 60mg Tab
- RT1T2 (Experimental): Period I: R, "Lixiana 60mg" with 150mL water Period II: T1, "DA-5209 60mg" without water Period III: T2, "DA-5209 60mg" with 150mL water
  Interventions: Drug: DA-5209 60mg Tab; Drug: Lixiana 60mg Tab
- RT2T1 (Experimental): Period I: R, "Lixiana 60mg" with 150mL water Period II: T2, "DA-5209 60mg" with 150mL water Period III: T1, "DA-5209 60mg" without water
  Interventions: Drug: DA-5209 60mg Tab; Drug: Lixiana 60mg Tab
- T2RT1 (Experimental): Period I: T2, "DA-5209 60mg" with 150mL water Period II: R, "Lixiana 60mg" with 150mL water Period III: T1, "DA-5209 60mg" without water
  Interventions: Drug: DA-5209 60mg Tab; Drug: Lixiana 60mg Tab
- T2T1R (Experimental): Period I: T2, "DA-5209 60mg" with 150mL water Period II: T1, "DA-5209 60mg" without water Period III: R, "Lixiana 60mg" with 150mL water
  Interventions: Drug: DA-5209 60mg Tab; Drug: Lixiana 60mg Tab

INTERVENTIONS:
Drug: DA-5209 60mg Tab — single oral administration of 1 tablet of "DA-5209 60mg Tab" with 150mL water
Drug: DA-5209 60mg Tab — single oral administration of 1 tablet of "DA-5209 60mg Tab" without water
Drug: Lixiana 60mg Tab — single oral administration of 1 tablet of "Lixiana 60mg Tab" with 150mL water

SUMMARY:
An Open-Label, Randomized, 6-sequence, 3-period, Fasting Condition, Single-dose, Per Oral, Cross-over Study to Evaluate the Bioequivalence between "DA-5209 60mg Tab" and "Lixiana 60mg Tab" in Healthy Volunteers

DETAILED DESCRIPTION:
1. Study design: An open-Label, randomized, 6-sequence, 3-period, fasting condition, single-dose, per oral, cross-over study
2. Administration method:

   The subject should maintain a minimum of 10 hours of empty stomach before administration, and give an oral dose of 1 tablets (DA-5209 60mg) without water or (DA-5209 60mg or Lixiana 60mg) with 150 mL of water at around 8 a.m. on the day of the test. The subject should not chew or break the drug, but should swallow in whole with water. The difference in administration time between the test subjects is about one minute apart, considering the blood collection time.
3. Wash out period: at least 7 days
4. Blood collection time: Before the administration, 5, 10, 15, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hr after the administration (total 15 times)
5. Analysis: Measurement of the concentration of an unchangeable substance of Edoxaban in plasma

ELIGIBILITY:
Inclusion Criteria:

1. A person who aged 19 or older at the time of screening
2. BMI of 18 to 30 (BMI calculation: kg/m2)

   ◦Males or Females weighing 60kg or more
3. No congenital or chronic diseases or pathological symptoms
4. A person who is judged to be suitable for the study by the investigator based on the clinical laboratory examination
5. A person who has fully understood the contents of the consent form for the study and signed the consent form voluntarily and recorded the date of signature
6. A person who agreed to use contraception from the first administration of IP to a week after the last administration of IP

Exclusion Criteria:

1. A person who has taken a drug that significantly induces (e.g., barbital) or inhibits the drug metabolic enzyme within 30 days prior to the first administration of IP
2. A person who has participated in other clinical trials within six months prior to the first administration of the IP
3. A person who has had whole blood transfusion within 2 months or the apheresis within 2 weeks before the first administration of IP
4. A person who has medical history of gastric resection that can affect the drug absorption
5. A person with a history of regular alcohol intake within a month prior to the first administration of the IP:

   * Male: More than 21 cups/week
   * Female: More than 14 cups/week (1 cup: 50 ml of soju, 250 ml of beer, 30ml of spirits)
6. A person who is hypersensitive to any of the IP components, with clinically significant bleeding, with end-stage renal disease and have kidney dialysis, with hepatic disease related to blood coagulation disorder and clinically significant risk of bleeding, with severe liver impairment, with an increased risk of bleeding, use combination therapy with other anticoagulants, Severe hypertension factor, have undergone artificial heart valve replacement
7. A person who has medical history of mental disease
8. A person who is judged not to be suitable for the study by the investigator
9. Lactating or possibly pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Area Under the plasma Concetration versus time curve(AUCt) of Edoxaban | Before administration ~ 48hours
  Area Under the plasma Concetration versus time curve(AUCt) of Edoxaban
Peak Plasma Concentration(Cmax) of Edoxaban | Before administration ~ 48hours
  Peak Plasma Concentration(Cmax) of Edoxaban

SECONDARY OUTCOMES:
Absorption rate constant(Ka) of Edoxaban | Before administration ~ 48hours
  Absorption rate constant(Ka) of Edoxaban
% of concentration compared to Maximum observed plasma concentration(Cmax) of Edoxaban | Before administration ~ 48hours
  % of concentration compared to Maximum observed plasma concentration(Cmax) of Edoxaban
Area under the plasma drug concentration-time curve from time 0 to infinity(AUC∞) of Edoxban | Before administration ~ 48hours
  Area under the plasma drug concentration-time curve from time 0 to infinity(AUC∞) of Edoxban
Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity(AUCt/AUC∞) of Edoxaban | Before administration ~ 48hours
  Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity(AUCt/AUC∞) of Edoxaban
Time of peak concentration(Tmax) of Edoxaban | Before administration ~ 48hours
  Time of peak concentration(Tmax) of Edoxaban
Terminal phase of Half-life(t1/2) of Edoxaban | Before administration ~ 48hours
  Terminal phase of Half-life(t1/2) of Edoxaban

CONTACTS AND LOCATIONS:
Overall Officials: SeungHyun Kang, Ph.D, Principal Investigator — H Plus Yangji Hospital
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea